CLINICAL TRIAL: NCT01633515
Title: Intralesional Cryosurgery for the Treatment of Basal Cell Carcinoma of the Lower Extremities in the Elderly - a Feasibility Study
Brief Title: Intralesional Cryosurgery for Basal Cell Carcinoma - a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Har-Shai, Head of plastic department, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMC-12-0032-CTIL
Record Dates: First submitted 2012-06-09; First posted 2012-07-04 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Basal Cell Carcinoma (BCC)
Keywords: Basal cell carcinoma (BCC); Cryotherapy; Cryosurgery
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intralesional cryotherapy (Other): 10 BCC (skin lesions) in the lower extremity of elderlies with risk factors for surgical complications.
  Interventions: Procedure: Intralesional cryotherapy

INTERVENTIONS:
Procedure: Intralesional cryotherapy — The Intralesional cryotherapy technology (CryoShape; CryoShape™, U.S Patent Number 6,503,246; European Patent Number 1299043, FDA 510(k) Number K060928) had been developed for the treatment of hypertrophic scars and keloids. The cryoneedle is connected by an adaptor to a cryogun filled with liquid nitrogen, and is introduced into the BCC. After the BCC is completely frozen, the cryoprobe defrosts and is withdrawn.
  Other relevant intervention: The cryotherapy will be performed under local anesthesia (bupivacaine). After the procedure topical antibiotic cream will be applied. Participants will be followed at the out patient clinic for an average duration of 5 month after cryotherapy (3 month post cyotherapy until the biopsy and then 1-2 month more until biopsy results are received).
  Other Names: CryoShape; CryoShape™, FDA 510(k) Number K060928)

SUMMARY:
A feasibility study for the treatment of Basal Cell Carcinoma of the lower extremities in the elderly utilizing intralesional cryosurgery.

10 cases of BCC (confirmed by biopsy) in the lower extremity of elderly will undergo intralesional cryotherapy. A Cryoneedle is introduced through the skin lesion (BCC) and thus the BCC is frozen. Treatment success will be determined according to biopsy results 3 months after treatment

DETAILED DESCRIPTION:
BCC is the most common skin cancer. Many treatment modalities are acceptable including cryotherapy - freezing of the skin lesion with liquid nitrogen. This method is highly effective for the treatment of BCC. The purpose of this study is to determine the cure rates of BCC utilizing intralesional cryotherapy.

surgery in the gold standard for the treatment of BCC, however in the case of skin malignancy in the elderly and in the lower extremity, surgical complication (including skin grafting) are high. Therefore cryotherapy which is a non surgical treatment method provides an optimal therapeutic choice.

10 cases of BCC (confirmed by biopsy) in the lower extremity of elderly will undergo intralesional cryotherapy. A Cryoneedle is introduced through the skin lesion and the BCC is frozen. Treatment success will be determined according to biopsy results 3 months after treatment. Participants will be followed at the out patient clinic for the duration of wound healing, an expected average duration of 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 60 years old
* BCC was determined with tissue diagnosis in the lower extremity
* One or more risk factor for surgical complication including: diabetes, venous insufficiency, obesity, peripheral vascular disease, lymphedema and long term steroids use.

Exclusion Criteria:

* Patient unable to read, understand and sign the consent form

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Cure rate of intralesional cryotherapy for BCC in the lower extremity of elderly | Participants will be followed at the out patient clinic for an average duration of 5 month after cryotherapy (3 month post cyotherapy until the biopsy and then 1-2 month more until biopsy results are received).
  Cure rates of BCC in the lower extremity of elderly treated with intralesional cryotherapy. A biopsy will be performed 3 month post cryotherapy, the rate of biopsies which determine that no residual tumor is left will be defined as cure rate

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Har-Shai, M.D, Principal Investigator — Carmel Medical Center
Locations (1):
- Lin Medical Center, Haifa, Israel

REFERENCES:
- [Background] Har-Shai Y, Brown W, Pallua N, Zouboulis CC. Intralesional cryosurgery for the treatment of hypertrophic scars and keloids. Plast Reconstr Surg. 2010 Nov;126(5):1798-1800. doi: 10.1097/PRS.0b013e3181ef823d. No abstract available. PMID 21042160
- [Background] Har-Shai Y, Brown W, Labbe D, Dompmartin A, Goldine I, Gil T, Mettanes I, Pallua N. Intralesional cryosurgery for the treatment of hypertrophic scars and keloids following aesthetic surgery: the results of a prospective observational study. Int J Low Extrem Wounds. 2008 Sep;7(3):169-75. doi: 10.1177/1534734608322813. PMID 18757392
- [Background] Giuffrida TJ, Jimenez G, Nouri K. Histologic cure of basal cell carcinoma treated with cryosurgery. J Am Acad Dermatol. 2003 Sep;49(3):483-6. doi: 10.1067/s0190-9622(03)00903-4. PMID 12963913